CLINICAL TRIAL: NCT03373539
Title: Neurotrophin Expression in Infants as a Predictor of Respiratory and Neurodevelopmental Outcomes
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Fariba Rezaee, Staff, The Cleveland Clinic
Other Study IDs: 14-1270
Record Dates: First submitted 2017-12-08; First posted 2017-12-14 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2019-08

CONDITIONS: Bronchopulmonary Dysplasia; Chronic Lung Disease
Keywords: Biomarkers; Neurotrophins
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Important developmental processes continue until the completion of 40 weeks gestation. Even during fetal life, intrinsic and environmental factors determine the balance between health and the onset and development of diseases. Thus, it is crucial to understand the mechanisms that regulate normal development and the pathways that contribute to disease pathogenesis.

Neurotrophins are a family of four proteins that support the growth and survival of neurons. Their secretion increases during brain development, when new neurons are being formed and existing ones are branching to assemble complex neuronal circuits. In addition to their role in promoting neuron growth and development, neurotrophins are also a product of neuronal activity. Neurotrophins are also responsible for the maintenance of peripheral sensory neurons, including those in the lungs. Airway innervation is responsible for many aspects of lung function including the regulation of airway smooth muscle tone, mucus secretion, and reactivity; therefore, a physiological expression of neurotrophins in the lungs is required for normal lung function.

DETAILED DESCRIPTION:
Currently, there is no reliable method to identify infants who will have poor neurodevelopmental and respiratory outcomes. The ability to make such predictions would be beneficial for both making care decisions in the neonatal intensive care unit and for identifying infants who require earlier and more intense intervention. We intend to determine if neurotrophins can be utilized to predict an infant's long-term outcomes. Neurotrophins are a family of four proteins that support the growth and survival of neurons. Their levels have been shown to increase with brain development and decrease with brain injury. Neurotrophins have also been associated with development of airway injury in the neonate and later respiratory disease such as asthma. We plan to correlate serum neurotrophin levels with respiratory outcomes and neurological outcomes.

ELIGIBILITY:
Inclusion Criteria:

intubated infants in the Neonatal Intensive Care Unit (NICU)

Exclusion Criteria:

unwilling or unable to give or obtain informed consent

Ages: 1 Day to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: neonates in Neonatal Intensive Care Unit (NICU)
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Correlation of serum neurotrophins with development for Bronchopulmonary Dysplasia | within 48 hours of Neonatal Intensive Care Unit admission
  Neurotrophins include Nerve Growth Factor (NGF) and Brain-factor Neurotrophic Factor (BDNF)
Change in serum neurotrophins with developmental delays in children | Within 48 hours of Neonatal Intensive Care Unit admission, at 4 months, 1 year and 2 years
  Neurotrophins include Nerve Growth Factor (NGF) and Brain-factor Neurotrophic Factor (BDNF)
Change in serum neurotrophins with respiratory outcomes in children | Within 48 hours of Neonatal Intensive Care Unit admission, at 4 months, 1 year and 2 years
  Neurotrophins include Nerve Growth Factor (NGF) and Brain-factor Neurotrophic Factor (BDNF)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Piedimonte, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States